CLINICAL TRIAL: NCT04182802
Title: Using Benralizumab to Explore Treatment Response Patterns in Functional Lung MRI and Advanced Measures of Lung Function
Brief Title: MRI and Lung Function Measures of Benralizumab Response in Asthma
Acronym: MR BEN
Status: Withdrawn | Type: Observational
Why Stopped: Funding withdrawn due to COVID related delays.
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); University of Sheffield (Other); University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: STH20679
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- eosinophilic asthma

SUMMARY:
New treatments have been developed for asthma that are good at preventing asthma attacks and improving day-to-day symptoms. Alongside the development of these new drugs, there are new ways of measuring how the lung is affected by asthma. In particular, investigators have developed ways of seeing how air moves in the lungs of people with asthma, using MRI scanning. This study aims to see how quickly these new drugs result in changes in the way the lung is working, as seen in the MRI scans and other breathing tests. This will help clinicians in the future to decide who is likely to respond to these new medicines, and once patients have started taking the drugs, will help clinicians to decide whether long term treatment is likely to benefit the people receiving them.

In this study, the investigators plan to do extra breathing tests and MRI scans on people who are receiving the drug as part of their usual clinical care. The study will not change an individual's treatment, but will give the investigators more information about the patients' illnesses and the way the patients' bodies respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

* People with eosinophilic asthma meeting the National Institute for Health and Clinical Excellence (NICE) criteria for benralizumab therapy based on eosinophil count and exacerbation rates will be offered the chance to participate in this study.

Exclusion Criteria:

* Any medical illness that in the opinion of the investigator is likely to significantly impact on the response to benralizumab or the outcome of the MRI and lung function testing.
* Non-concordance with routine asthma therapies (this would be assessed as a mandatory part of NICE-based criteria).
* Any additional significant lung illness that would impact on likelihood of response to benralizumab. Of note, trivial stable bronchiectasis that in the opinion of the patient's clinician is not clinically significant nor likely to result in either recurrent exacerbations or impairment of interpretation of investigation results will not be exclusion criteria. Part of the initial inclusion regarding eligibility by NICE criteria include an assessment of a likely eosinophilic asthmatic phenotype with probability of treatment response, and potential subjects with complex lung disease would be unlikely to be eligible.
* Current cigarette smoking, or cigarette smoking within the past 6 months
* Significant lifetime smoking history of ≥20 pack years
* Previous use of another biologic therapy targeting eosinophils within 6 months of enrollment
* Pregnancy, planning pregnancy, or breast feeding. Women of childbearing potential must use effective contraception (concordant use of hormonal contraceptive, intrauterine device, total abstinence), and urine pregnancy tests will be performed before scans.
* Abnormal renal function (eGFR <30), to avoid risks from Gadolinium chelate MRI contrast agents.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a pragmatic, cohort feasibility study, the primary aim of which is to determine which parameters of functional and structural lung MRI change over what time course after the introduction of a anti-eosinophil strategy in people with eosinophilic asthma.
  At present, the first-line licensed choice for anti-eosinophil therapies is mepolizumab, which has been shown to be effective at reducing exacerbations of asthma. Mepolizumab is given every 4 weeks. Benralizumab has two possible advantages over mepolizumab: swifter onset, and less frequent administration (it is given 4 weekly for the first three injections, then 8 weekly). People who would be eligible for either therapy will be offered a choice of participating in this clinical study or receiving mepolizumab through standard NHS pathways.
  Candidate patients will be identified in severe asthma clinics at Sheffield Teaching Hospitals and through the associated clinics at Rotherham, Doncaster, Barnsley and Chesterfield.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-13 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage ventilated lung volume | Baseline to 16 weeks
  Measurement of lung volume assessed by magnetic resonance imaging

IPD SHARING:
Plan to Share IPD: Undecided